CLINICAL TRIAL: NCT03586453
Title: A Phase II Study of Osimertinib With On-study and Post-progression Biopsy in the First Line Treatment of EGFR Inhibitor naïve Advanced EGFR Mutant Lung Cancer
Brief Title: Osimertinib In EGFR Mutant Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Pasi Janne, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-070
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Cell Lung Cancer (NSCLC); Epidermal Growth Factor Receptor (EGFR) mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Osimertinib (Experimental): Osimertinib: Oral, once a day, dosage determined per protocol
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Patients who fulfill eligibility criteria will be entered into the trial to receive Osimertinib.
  After the screening procedures confirm participation in the research study:
  * Osimertinib: Oral, Daily 28 day cycle.
  * Radiographic assessment: every 2 cycles for first 6 months and then every 3 cycles until disease progression.
  * Tumor biopsy between C4 and C8 and at disease progression
  Other Names: Tagrisso; AZD9291

SUMMARY:
This research study is studying a targeted therapy as a possible treatment for Non-Small Cell Lung Cancer (NSCLC) with an EGFR mutation.

The names of the study drug involved in this study is:

- Osimertinib (Tagrisso)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

This research study is studying a targeted therapy as a possible treatment for Non-Small Cell Lung Cancer (NSCLC) with an EGFR (epidermal growth factor receptor) genetic mutation. The EGFR gene produces a protein that helps cells divide. Specific changes or a mutation in the genetic information causes abnormal cell division and can lead to lung cancer. Patients who have NSCLC with an EGFR gene mutation can be treated by drugs called EGFR tyrosine kinase inhibitors (EGFR TKIs). They may stop (or "inhibit") the effect of the mutation in the EGFR gene.

- Osimertinib has been approved by the FDA (the U.S. Food and Drug Administration) for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed stage IV NSCLC (per AJCC 7th edition) with either the L858R or exon 19 deletion activating EGFR mutation as identified in a CLIA-approved laboratory from tumor tissue.

  --Note: recurrent stage IV disease initially diagnosed at an earlier stage is considered eligible, provided prior treatment criteria is met.
* Participants must have measurable disease at baseline, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Participants must be aged ≥ 18 years
* Participants must have an ECOG performance status of 0-1 (Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * hemoglobin >9.0 g/dL
  * total bilirubin < 1.5 times the ULN if no liver metastases or < 3 times the ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases
  * AST(SGOT)/ALT(SGPT) <2.5 × institutional upper limit of normal or <5 times the ULN in the presence of liver metastases
  * creatinine ≤ 1.5 x institutional upper limit of normal

    --- OR
  * creatinine clearance ≥50 mL/min as determined by the Cockcroft-Gault formula.
  * Note: For participants entering study after starting commercial osimertinib, elevations in hepatic transaminases (AST/ALT) and/or total bilirubin < grade 2 at study entry are acceptable (see protocol Table 2).
* Participants must have biopsy tissue at time of diagnosis available and sufficient for targeted next-generation sequencing. The sequencing can be performed at a commercial vendor such as Foundation Medicine. The testing does not have to be completed prior to study enrollment. If the specimen is insufficient a repeat biopsy will need to be performed.

  --Note: Cytology specimen may be acceptable for baseline NGS if tumor cellular content is sufficient and following PI approval. If there is no cytology specimen or tissue sample available for NGS, plasma-based NGS may be acceptable for enrollment following discussion with PI.
* For participants entering study after starting commercial osimertinib: a tissue sample from the time of diagnosis must be available and sufficient for NGS testing. Participants who have had commercial tumor NGS testing performed on their pre-osimertinib treated specimen do not need NGS repeated as part of this study.
* Participants must be willing to undergo a repeat tumor biopsy during study treatment between cycles 4 and 8 (if considered medically safe) and at the time of disease progression.
* Participants must be ≥2 weeks since any major surgery (excluding vascular access placement, mediastinoscopy, or biopsies performed by an interventional service)
* Male patients should be asked to use barrier contraceptives (i.e., by use of condoms) during sex with all partners who are women of child bearing potential, including pregnant women, during the trial and for a washout period of 4 months. Male patients should avoid procreation for 4 months after completion of trial treatment. Patients should refrain from donating sperm from the start of dosing until 4 months after discontinuing study treatment.
* Female patients (women of child-bearing potential): Willing to use adequate contraception (barrier or abstinence) at least 2 weeks before receiving any study medication, while on treatment with study drug, and for 6 weeks after finishing treatment.
* Female patients: Must not be pregnant or breast-feeding. Women of child-bearing potential must have a negative pregnancy test (urine or serum) prior to start of dosing or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * a) Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
  * b) Women under 50 years are considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution.
  * c) Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.
* Ability to understand and the willingness to sign a written informed consent document.
* Subjects may enter the study even if they have started their treatment using commercial osimertinib. Subjects may enter the study anytime during the first 3 months of receiving commercial osimertinib therapy (up to 84 days of commercial osimertinib before entering the study). In order to enter the study after starting commercial osimertinib, subjects must meet all eligibility criteria listed above, have baseline and follow up imaging available for review for response assessment, and must not have developed disease progression during the first 3 months of commercial osimertinib therapy.

Exclusion Criteria:

* Subjects should not enter the study if any of the following exclusion criteria are fulfilled:
* Prior or ongoing treatment with any of the following:

  * EGFR targeted therapy (TKI or antibody) or any other targeted therapies targeting the ERBB family except for subjects receiving first line osimertinib during the first three months of therapy.
  * Any cytotoxic chemotherapy, investigational agents, immunotherapy or anticancer drugs for the treatment of metastatic NSCLC
  * Note: Patients who have completed adjuvant or neo-adjuvant chemotherapy > 6 months ago are considered treatment naïve
* Prior radiotherapy, including CNS radiation, within 2 weeks of the first dose of study treatment.
* Uncontrolled central nervous system (CNS) disease, including parenchymal brain metastases, leptomeningeal disease, or spinal cord compression. Patients with asymptomatic untreated brain metastases are eligible. Patients with treated CNS disease will be allowed to enroll provided they have asymptomatic clinically confirmed stable disease with ≥2 weeks since definitive CNS therapy (radiation or surgery) and ≥2 weeks without systemic steroids. Patients may undergo either whole brain radiation or stereotactic radiosurgery prior to study entry.
* History of allergic reactions attributed to compounds, or any of its excipients, of similar chemical or biologic composition to osimertinib.
* Patients currently receiving and unable to stop using medications or herbal supplements known to be potent inhibitors or inducers of CYP3A4. The full list of medications that would make a patient ineligible are provided in Appendix B, along with indicated washout times.
* Any unresolved toxicities from prior therapy, including commercial osimertinib, greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment.
* Malignancies within the past 3 years excluding adequately treated basal or squamous cell carcinomas of the skin without local or distant metastases.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, previous significant bowel resection, or any process that compromises the ability to swallow or absorb oral medication
* Significant medical history or unstable medical comorbidities, including:

  * heart disease including congestive heart failure (NYHA Grade II or greater); unstable angina; prior myocardial infarction (NSTEMI or STEMI) within 6 months prior to study enrollment; hypertension with a systolic blood pressure of >150 mm Hg or diastolic blood pressure of >100 mm Hg while on antihypertensive medication
  * any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, e.g. complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250msec, have normal QT interval on ECG evaluation QT corrected Fridericia (QTcF) of ≤ 450 ms in males or ≤ 470 ms in females
  * any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives, or any concomitant medication known to the prolong the QT interval and cause Torsades de Pointes and listed in Appendix B that a patient is unable to stop
  * past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
  * active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol
  * known active infection or ongoing antiviral medication for viral infections including hepatitis B, hepatitis C, or human immunodeficiency virus (HIV). Screening for chronic conditions is not required. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with osimertinib.
  * cardiac ejection fraction of < 45%
  * Any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol
* Known to be T790M+ (on pre-treatment tumor or plasma) or known germline T790M. Note: testing is not required for study entry.
* Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry. Women of child-bearing potential must have a negative pregnancy test prior to start of dosing.
* Pregnant women are excluded from this study because the effects of osimertinib on the development of the fetus are unknown, and there is potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with osimertinib, breastfeeding should be discontinued if the mother is treated with osimertinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Mechanisms of resistance to Osimertinib | 4 Months
  Evaluated by comparing the genomic changes using targeted next generation sequencing in the post-osimertinib tumor to the pre-treatment tumor specimen.

SECONDARY OUTCOMES:
Best objective response | 6 months
  Best objective response will be evaluated via RECIST 1.1 criteria. RECIST1.1 measurements of CT scans will be measured every 2 cycles on treatment to determine the objective response rate for patients being treated with osimertinib.
Overall Response Rate | 3 years
  Defined as the proportion of patients with best response of CR or PR per investigator assessment using RECIST 1.1. start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started.
Progression-free survival (PFS) | 2 years
  Time from registration to documented disease progression or death from any cause, whichever occurs first. The Kaplan-Meier method will be used to determine the progression-free survival of patients enrolled on protocol and treated with combination osimertinib and selumetinib.
Overall survival | 2 years
  Survival follow-up with clinic visits or phone calls will be used to monitor for overall survival from time of study randomization to death from any cause. The Kaplan-Meier method will be used to calculate overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A Jänne, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No